CLINICAL TRIAL: NCT07299136
Title: Evaluating the Effect of Hugging and Praying on Traumatic Birth Perception, Birth Pain, and Birth Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: nurten özçalkap (Other)
Collaborators: Agri Ibrahim Cecen University (Other)
Responsible Party: Sponsor-Investigator, nurten özçalkap, Asistant Professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/38
Record Dates: First submitted 2025-11-28; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: The Effect of Hugging and Praying on Traumatic Birth Perception, Pain, and Anxiety
Keywords: birth; hugging; praying; pain; anxiety; trauma
MeSH Terms: conditions — Pain; Anxiety Disorders; Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Hugging
  Interventions: Other: Hugging group,
- Group 2 (Experimental): Praying
  Interventions: Other: Prayer group
- Group 3 (Experimental): Hugging and Praying
  Interventions: Other: Hugging and Praying group
- Group 4 (No Intervention): CONTROL

INTERVENTIONS:
Other: Hugging group, — For the hugging group, hugging sessions will be provided whenever the pregnant woman desires and during contractions, if she wishes, by a close relative (husband, mother, sister, etc.) or midwife. The pregnant woman can be hugged for as long as she wants or for 5-10 minutes.
  Arms: Group 1
Other: Prayer group — For the prayer group, whenever the pregnant woman wishes, or during contractions if she wishes, a close relative (husband, mother, sister, etc.) or midwife will recite a prayer of the pregnant woman's choice, if she has one; if she does not have a preferred prayer, the first 5 verses of Surah Al-Inshiqaq will be recited:
  In the name of Allah, the Most Gracious, the Most Merciful
  1. When the sky is split asunder,
  2. And obeys the command of its Lord,
  3. When the earth is stretched out flat,
  4. And casts forth what is within it,
  5. And obeys the command of its Lord, every person will be confronted with what they have done! To be recited together
  Arms: Group 2
Other: Hugging and Praying group — The Hugging and Praying group will perform both hugging and praying together with the woman.
  Arms: Group 3

SUMMARY:
Pregnant women participating in our study will receive the intervention (hugging, praying, and hugging + praying) from the researcher or a relative as often as they wish during labor and contractions. These sessions will be administered during each stage of labor, taking into account when the pregnant woman is ready to begin the intervention.

DETAILED DESCRIPTION:
Pregnant women participating in our study will receive the intervention (hugging, praying, and hugging + praying) from the researcher or a relative as often as they wish during labor and contractions. These sessions will be administered during each stage of labor, taking into account when the pregnant woman is ready to begin the intervention.

For the hugging group, hugging sessions will be performed whenever the pregnant woman wants and during contractions, if she wishes, by a relative (husband, mother, sister, etc.) or midwife. The pregnant woman can be hugged for as long as she wants or for 5-10 minutes. For the prayer group, whenever the pregnant woman wishes, or during contractions if she wishes, a close relative (husband, mother, sister, etc.) or midwife will recite a prayer chosen by the pregnant woman, if she has one; if she does not have a preferred prayer, the first 5 verses of Surah Al-Inshiqaq will be recited:

In the name of Allah, the Most Gracious, the Most Merciful

1. When the sky is split asunder,
2. And obeys the command of its Lord,
3. When the earth is stretched out flat,
4. And casts forth what is within it,
5. And obeys the command of its Lord, every person will be confronted with what they have done! To be read together Before starting the first session, the "Information Form," "Visual Analog Scale," Traumatic Birth Perception Scale, and "Oxford Birth Anxiety Scale (Appendix 4)" will be administered. and at the end of the first, second, and fourth stages of birth, the "Visual Analog Scale," "Traumatic Birth Perception Scale," and "Oxford Birth Anxiety Scale" will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years

  * No communication barriers
  * Applying to Ağrı Training and Research Hospital for normal delivery within the study dates
  * Volunteering to participate in the study
  * No contraindications for normal vaginal delivery (e.g., cephalopelvic disproportion)
  * Being at term (38-42 weeks)
  * No condition preventing praying and hugging

Exclusion Criteria:

* Refusal to participate in the study
* Maternal disease (heart disease, diabetes, etc.)
* Having a preterm or postterm pregnancy
* Undergoing an emergency cesarean section during follow-up
* Having a fetal malformation (anencephaly, Down syndrome, etc.)
* Not answering the questions in the questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 164 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Information Form | Before starting the first session average 8 months
  This form, prepared by the researcher in line with the literature, inquires about the socio-demographic characteristics of the participants.
Visual Analog Scale (VAS) | average 8 months
  It is a one-dimensional scale that objectively assesses a pregnant woman's perception of pain. It allows some values that cannot be measured numerically to be converted into numerical values. In 1921, Hayes and Peterson argued that emotional levels could be expressed on lines. The VAS was first developed and used by Bond and Pilowsky in 1966. The VAS is a 100 mm (10 cm) ruler used to quantitatively determine pain intensity, with one end representing painlessness (0 = no pain) and the other end representing the most severe pain (10 = severe pain). The patient marks any point between the two points that corresponds to the severity of their pain. The distance between the end of the scale representing painlessness and the point marked by the patient is measured with a ruler and recorded in centimeters. This numerical value indicates the pregnant woman's pain intensity. 0 cm = No pain, 0.53 cm = Mild pain, 3.5-6.5 = Moderate (Ergin, 2013; Aslan, 2006; Mucuk, 2009).
Traumatic Birth Perception Scale | average 8 months
  TThe Traumatic Birth Perception Scale (TBRS), developed by Yalnız et al. in 2016, is a thirteen-item, unidimensional Likert-type separation scale (Yalnız et al., 2016). Scores range from 0 to 10 for all items not requiring reverse scoring. The minimum scale score is 0 and the maximum is 130. The total scale score ranges from 0 to 26, indicating very low levels of perception of traumatic birth; 27 to 52, indicating low levels; 53 to 78, indicating moderate levels; 79 to 104, indicating high levels; and 105 to 130, indicating very high levels of perception of traumatic birth. The scale's Cronbach's alpha coefficient is .89 (Yalnız et al., 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Özçalkap, Principal Investigator — AĞRI İBRAHİM ÇEÇEN UNIVERSTY; SİBEL YÜCETÜRK, Asist. Prof., Study Chair — SİNOP UNIVERSTY; AYŞE Çuvadar, Assot Prof., Study Director — KARABUK UNIVERTY
Locations (1):
- Ağri İbrahim Çeçen Universty, Ağrı, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we don't share individual participant data with other researchers

REFERENCES:
- [Result] Redshaw M, Martin C, Rowe R, Hockley C. The Oxford Worries about Labour Scale: women's experience and measurement characteristics of a measure of maternal concern about labour and birth. Psychol Health Med. 2009 May;14(3):354-66. doi: 10.1080/13548500802707159. PMID 19444713